CLINICAL TRIAL: NCT03422029
Title: Study to Evaluate the Efficacy and Safety of 177Lu-Dotatate PRRT in Metastatic GEP-NEN Patients
Brief Title: Efficacy and Safety of 177Lu-Dotatate PRRT in Metastatic GEP-NEN Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Shen Lin, MD, Professor, Chief of Department of GI Oncology, Peking University Cancer Hospital, Peking University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRRT
Record Dates: First submitted 2018-01-30; First posted 2018-02-05 (Actual); Last update posted 2020-02-07 (Actual); Status verified 2020-02

CONDITIONS: Neuroendocrine Tumors
Keywords: ORR; Safety; PFS
MeSH Terms: conditions — Neuroendocrine Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 177Lu-Dotatate PRRT (Experimental): 177Lu-Dotatate A maximum of 8 cycles of 1000mCi 177Lu-Dotatate, each. Route of administration: Slow intravenous infusion/injection (i.v.) Duration of treatment: 8 cycles, every 8 weeks
  Interventions: Drug: 177Lu-Dotatate PRRT

INTERVENTIONS:
Drug: 177Lu-Dotatate PRRT — PRRT using 177Lu-Dotatate 100-150mCi will be performed 8-weekly. A maximum of 8 cycles will be administered.
  Other: Amino-Acid Solution The Amino-Acid Solution (AAS) to be used in this study, infused over 4-6 h, starting 30 min before PRRT

SUMMARY:
The purpose of the study is to evaluate efficacy and safety of Peptide Receptor Radionuclide Therapy (PRRT) with 177Lu-Dotatate in patients with inoperable, progressive, somatostatin receptor-positive (SSTR+), neuroendocrine tumours of GEP-NEN

ELIGIBILITY:
Inclusion Criteria:

1. sign written informed consent form
2. age ≥ 18 years
3. pathologically confirmed well-differentiated neuroendocrine tumors;
4. unresectable metastatic tumors confirmed by radiological imaging;
5. Somatostatin receptor positive (SSTR+) disease;
6. Radiological disease progression within 12 months, defined as progressive disease per RECIST 1.1. criteria
7. No more than 2 prior antitumor drugs, including somatostatin analogs, targeted drugs and chemotherapy, with the last dose over 4 weeks;
8. At least 1 measurable lesion (only 1 measurable lymph node lesion is excluded) (routine CT scan >=20mm, spiral CT scan >=10mm, no prior radiation to measurable lesions);
9. Screening laboratory values must meet the following criteria (within past 7 days): hemoglobin ≥ 9.0 g/dL; neutrophils ≥ 1500 cells/ μL; platelets ≥ 100 x 10^3/ μL; total bilirubin ≤ 1.5 x upper limit of normal (ULN); aspartic transaminase (AST) and alanine transaminase (ALT) ≤ 2.5 x ULN without, and ≤ 5 x ULN with hepatic metastasis; serum creatinine ≤1╳ULN;
10. KPS ≥ 70;
11. Predicted survival >=3 months;
12. Negative serum or urine pregnant test within 7 days prior to randomization for child-bearing age women;
13. Sexually active males or females willing to practice contraception during the study until 30 days after end of study.

Exclusion Criteria:

1. Hypersensitivity to DOTA, lutetium-177, or any excipient of edotreotide or everolimus or any other Rapamycin derivative;
2. Prior antitumor therapy (including corticosteroids and immunotherapy) or participation in other clinical trials within past 4 weeks, or have not recovered from toxicities since the last treatment;
3. Received surgery within past 4 weeks, or have not recovered from surgery;
4. Concurrent severe infection；
5. Severe, uncontrolled medical condition that would affect patients' compliance or obscure the interpretation of toxicity determination or adverse events, including severe liver disease (active hepatitis, cirrhosis), uncontrolled diabetes or hypertension, or pulmonary disease ( interstitial pneumonia, obstructive pulmonary disease or symptomatic bronchospasm);
6. Prior long term steroid therapy (excluding short term steroid treatment which is completed prior to > 2 weeks of study enrollment)；
7. Meningeal carcinomatosis;
8. Patients with central nervous system(CNS) disorder or peripheral nervous system disorder or psychiatric disease；
9. Known history of uncontrolled or symptomatic angina, uncontrolled arrhythmias and hypertension, or congestive heart failure, or cardiac infarction within 6 months prior to study enrollment, or cardiac insufficiency；
10. Pregnant or nursing, or sexually active males or females refuse to practice contraception during the study until 30 days after end of study;
11. History of other malignancy. However, subjects who have been disease-free for 5 years, or subjects with a history of completely resected non-melanoma skin cancer or successfully treated in situ carcinoma, are eligible；
12. Person with no capacity (legally) or inappropriate to continue study treatment for ethics/medical reasons；
13. Underlying medical condition that, in the Investigator's opinion, would increase the risks of study drug administration or obscure the interpretation of toxicity determination or adverse events.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 20 (Estimated)
Dates: Start 2018-01-31 (Actual); Primary Completion 2020-12-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | From date of first dose until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  CT/MRI will be performed every 8 weeks for efficacy evaluation by RECIST 1.1 and CHOI
Incidence of Treatment-related Adverse Events（Safety and Tolerability） | From date of first dose until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0

SECONDARY OUTCOMES:
Progression-free survival | baseline, every 8 weeks up to 1 year after last patient first treatment
  Progression-free survival is defined as the time from the date of first dose to the date of the first documented radiological progression or death due to any cause

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No